CLINICAL TRIAL: NCT05303935
Title: Effects of Quetiapine on Sleep and Next Day Alertness in People With Obstructive Sleep Apnea
Acronym: QOSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Flinders University (Other)
Responsible Party: Principal Investigator, Professor Danny Eckert, Director, Adelaide Institute for Sleep Health, Flinders University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 4965
Record Dates: First submitted 2022-02-24; First posted 2022-03-31 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep apnea, obstructive; quetiapine; randomised; double-blind; placebo; respiratory arousal threshold
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Quetiapine Fumarate; Sugars

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled, cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quetiapine (Experimental): Quetiapine 50mg in the form of one capsule, taken before bedtime. Dosage is taken on one instance for one night only.
  Interventions: Drug: Quetiapine 50 MG
- Placebo (Placebo Comparator): Placebo sugar pill in the form of one capsule, taken before bedtime. Dosage is taken on one instance for one night only.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine 50 MG — A single dose of 50mg of quetiapine taken at bedtime for one night.
  Other Names: Seroquel
  Arms: Quetiapine
Drug: Placebo — A placebo sugar pill that looks like the quetiapine tablet taken at bedtime for one night.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Quetiapine is medication used to treat schizophrenia and bipolar disorder. Increasingly, low doses of quetiapine are prescribed "off-label" for insomnia. Quetiapine increases sleep duration with fewer interruptions, and people report feeling more rested. This accounts for why it is popular to prescribe for insomnia. Insomnia and obstructive sleep apnea (OSA) share many symptoms and differential diagnosis can be difficult. While quetiapine may improve sleep and breathing in certain people (i.e in light sleepers) an initial study indicated that quetiapine caused breathing disturbances in healthy individuals. Effects in OSA are unknown. In this placebo-controlled double blind study, participants with mild-moderate OSA will spend 2 nights in the sleep lab, one with quetiapine at a dose commonly prescribed for insomnia and one with placebo. The investigators will assess participants sleep by standard clinical sleep study, and morning alertness using questionnaires, reaction tests, and a driving simulator test.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 18+ (Adult, Older Adult)
* Gender: All
* Moderate or more "difficulty staying asleep" score on the Insomnia Severity Index questionnaire
* Obstructive Sleep Apnoea (OSA), Apnoea Hypopnea Index ≥ 5 events/hour
* BMI between 18.5 and 40 kg/m2

Exclusion Criteria:

* Concomitant medications that interact or are contraindicated with quetiapine
* Concomitant medications known to influence breathing, sleep, arousal, or muscle physiology
* Current pregnancy or breast-feeding
* Current or recent other medical conditions likely to affect results or safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Change in OSA severity (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  OSA severity as measured by the AHI (apnoea hypopnea index measured as # events/h sleep) during overnight in-laboratory polysomnography.

SECONDARY OUTCOMES:
Change in nadir overnight hypoxemia (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Nadir overnight oxygen saturation during sleep (%) measured via pulse oximetry during overnight in-laboratory polysomnography.
Change in mean overnight hypoxemia (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Mean overnight oxygen saturation during sleep (%) measured via pulse oximetry during overnight in-laboratory polysomnography.
Change in time below 90% blood arterial oxygen saturation (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Percent time asleep spent below an arterial oxygen saturation of 90% measured via pulse oximetry during overnight in-laboratory polysomnography.
Change in sleep efficiency (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Percent time spent asleep divided by the recording time from lights out to lights on during overnight in-laboratory polysomnography.
Change in arousal index (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Number of cortical arousals per hour of sleep during overnight in-laboratory polysomnography.
Change in sleep architecture (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Proportion of sleep stages (% total sleep time) during overnight in-laboratory polysomnography.
Change in respiratory control (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Loop gain and the ventilatory response to arousal (% eupnea) during overnight in-laboratory polysomnography.
Change in the respiratory arousal threshold (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Threshold to arousal (% eupnea) during overnight in-laboratory polysomnography.
Change in airway collapsibility (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Vpassive (% eupnea) during overnight in-laboratory polysomnography.
Change in pharyngeal muscle response (Quetiapine night vs. placebo night) | Two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Vcompensation (% eupnea) during overnight in-laboratory polysomnography.
Baseline OSA endotypes (outcomes 8-11) and whether they are associated with changes in OSA severity (Quetiapine night vs. placebo night) | Baseline sleep study
  Exploratory analysis to determine if baseline OSA endotypes (outcomes 8-11) are associated with changes in OSA severity (Quetiapine night vs. placebo night)
Change in perceived sleepiness (Quetiapine night vs. placebo night) | Next morning following two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Next day perceived sleepiness assessed via the Karolinska Sleepiness Scale (10 point scale where 1=extremely alert and 10=extremely sleepy)
Change in driving simulator performance (Quetiapine night vs. placebo night) | Next morning following two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Next day alertness as measured via the AusEd driving simulator performance task
Change in psycho-motor vigilance (Quetiapine night vs. placebo night) | Next morning following two non-consecutive single night sleep studies (Quetiapine night vs. placebo night) up to one month apart.
  Next day alertness as measured via the pschomotor vigilance test (PVT)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Eckert, PhD, Principal Investigator — Flinders University
Locations (1):
- Adelaide Institute for Sleep Health, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Participants will be informed in plain language through the consent form that their deidentified data may be made available to other researchers. Deidentified participant data will only be shared with other researchers upon request to the chief investigator after study publication and subject to ethical approval.
Supporting Information: Study Protocol, ICF
Time Frame: At conclusion of study and related publications.
Access Criteria: IPD may be shared for research purposes on application to the chief investigator and subject to applicable ethical review.

REFERENCES:
- [Background] Debernard KAB, Frost J, Roland PH. Quetiapine is not a sleeping pill. Tidsskr Nor Laegeforen. 2019 Sep 16;139(13). doi: 10.4045/tidsskr.19.0205. Print 2019 Sep 24. English, Norwegian. PMID 31556541
- [Background] McKean A, Monasterio E, Elliott T. How common is off-label prescription of quetiapine? N Z Med J. 2018 Oct 26;131(1484):77-78. No abstract available. PMID 30359361
- [Background] Pringsheim T, Gardner DM. Dispensed prescriptions for quetiapine and other second-generation antipsychotics in Canada from 2005 to 2012: a descriptive study. CMAJ Open. 2014 Oct 1;2(4):E225-32. doi: 10.9778/cmajo.20140009. eCollection 2014 Oct. PMID 25485247
- [Background] Cohrs S, Rodenbeck A, Guan Z, Pohlmann K, Jordan W, Meier A, Ruther E. Sleep-promoting properties of quetiapine in healthy subjects. Psychopharmacology (Berl). 2004 Jul;174(3):421-9. doi: 10.1007/s00213-003-1759-5. Epub 2004 Mar 17. PMID 15029469
- [Background] Karsten J, Hagenauw LA, Kamphuis J, Lancel M. Low doses of mirtazapine or quetiapine for transient insomnia: A randomised, double-blind, cross-over, placebo-controlled trial. J Psychopharmacol. 2017 Mar;31(3):327-337. doi: 10.1177/0269881116681399. Epub 2017 Jan 16. PMID 28093029
- [Background] Meira E Cruz M, Kryger MH, Morin CM, Palombini L, Salles C, Gozal D. Comorbid Insomnia and Sleep Apnea: mechanisms and implications of an underrecognized and misinterpreted sleep disorder. Sleep Med. 2021 Aug;84:283-288. doi: 10.1016/j.sleep.2021.05.043. Epub 2021 Jun 8. PMID 34214960
- [Background] Sweetman A, Lack L, McEvoy RD, Smith S, Eckert DJ, Osman A, Carberry JC, Wallace D, Nguyen PD, Catcheside P. Bi-directional relationships between co-morbid insomnia and sleep apnea (COMISA). Sleep Med Rev. 2021 Dec;60:101519. doi: 10.1016/j.smrv.2021.101519. Epub 2021 Jun 23. PMID 34229295
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Background] Eckert DJ. Phenotypic approaches to obstructive sleep apnoea - New pathways for targeted therapy. Sleep Med Rev. 2018 Feb;37:45-59. doi: 10.1016/j.smrv.2016.12.003. Epub 2016 Dec 18. PMID 28110857
- [Background] Eckert DJ, White DP, Jordan AS, Malhotra A, Wellman A. Defining phenotypic causes of obstructive sleep apnea. Identification of novel therapeutic targets. Am J Respir Crit Care Med. 2013 Oct 15;188(8):996-1004. doi: 10.1164/rccm.201303-0448OC. PMID 23721582
- [Background] Carter SG, Eckert DJ. Effects of hypnotics on obstructive sleep apnea endotypes and severity: Novel insights into pathophysiology and treatment. Sleep Med Rev. 2021 Aug;58:101492. doi: 10.1016/j.smrv.2021.101492. Epub 2021 Apr 22. PMID 33965721
- [Background] Eckert DJ, Owens RL, Kehlmann GB, Wellman A, Rahangdale S, Yim-Yeh S, White DP, Malhotra A. Eszopiclone increases the respiratory arousal threshold and lowers the apnoea/hypopnoea index in obstructive sleep apnoea patients with a low arousal threshold. Clin Sci (Lond). 2011 Jun;120(12):505-14. doi: 10.1042/CS20100588. PMID 21269278
- [Background] Khazaie H, Sharafkhaneh A, Khazaie S, Ghadami MR. A weight-independent association between atypical antipsychotic medications and obstructive sleep apnea. Sleep Breath. 2018 Mar;22(1):109-114. doi: 10.1007/s11325-017-1537-y. Epub 2017 Jul 13. PMID 28707161
- [Background] Sleep-related breathing disorders in adults: recommendations for syndrome definition and measurement techniques in clinical research. The Report of an American Academy of Sleep Medicine Task Force. Sleep. 1999 Aug 1;22(5):667-89. No abstract available. PMID 10450601
- See also: Compendium EM. SEROQUEL 25 mg film-coated tablets. 2021 [cited 2021 22/10/2021]. — http://www.medicines.org.uk/emc/product/5495/smpc
- See also: AstraZeneca. Australian Product Information Seroquel. 2020. — https://www.ebs.tga.gov.au/ebs/picmi/picmirepository.nsf/pdf?OpenAgent&id=CP-2020-PI-02417-1&d=20211103172310101